CLINICAL TRIAL: NCT06807814
Title: COMPERATIVE EFFECTS of CONSTRAINT- INDUCED MOVEMENT THERAPY and MIRROR THERAPY on FUNCTIONAL AMBULATION and QUALITY of LIFE in CHRONIC STROKE PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Mahrukh Syed, student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/246/08/24
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Stroke Rehabilitation; Mirror Therapy; Quality of Life (QOL)
Keywords: CONSTRAINT INDUCED MOVEMENT THERPHY; Stroke Rehabilitation; Mirror Therapy; Functional Ambulation; Quality Of Life
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: 1. Group A (Constraint-Induced Movement Therapy (CIMT
  2. Group B (Mirror Therapy):
Who Masked: Outcomes Assessor
Masking Description: Single-blinded assessor was considered to minimize bias in outcome measurements. The assessor was unaware of the intervention group assignment for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Constraint-Induced Movement Therapy (CIMT) (Experimental): A well-defined and structured rehabilitation program that restricts the use of the unaffected limb to promote the functional recovery of the affected limb in chronic stroke patients.
  Interventions: Combination Product: Constraint-Induced Movement Therapy (CIMT))
- Mirror Therapy (Experimental): A specific intervention that uses a mirror to create a visual illusion of the affected limb, with the goal of improving motor function and quality of life in chronic stroke patients.
  Interventions: Behavioral: Mirror Therapy

INTERVENTIONS:
Combination Product: Constraint-Induced Movement Therapy (CIMT)) — A well-defined and structured rehabilitation program that restricts the use of the unaffected limb to promote the functional recovery of the affected limb in chronic stroke patients(Franck et al., 2019). Sit-to-stand transitions, Indoor overground walking (forward, backward, and sideways), Weight-bearing movements in different directions: Stepping over obstacles and climbing stairs, Ideally, specific tasks to involve the paretic limb according to the activity of stroke survivors. This task was repeated ten times as part of the therapy sessions. Dynamic strengthening exercises like squats and lunges are integrated, progressively increasing intensity as patients gain confidence and strength. Balance and core stability exercises, including single-leg stances and seated weight shifts on therapy balls, address postural control and stability.(Cabanas-Valdés & Boix-Sala, 2021)
  Arms: Constraint-Induced Movement Therapy (CIMT)
Behavioral: Mirror Therapy — A specific intervention that uses a mirror to create a visual illusion of the affected limb, with the goal of improving motor function and quality of life in chronic stroke patients. The MT protocol included 10 minutes of warm-up, 1 hour of mirror box training, and 50 minutes of functional task practice. The warm-up activities included stretching and passive range of motion exercises. During the mirror box training, a mirror box that reflected the image of the unaffected arm was placed in the participant's midsagittal plane. Participants were required to symmetrically move both hands as simultaneously as possible while watching the reflection of the unaffected arm in the mirror as if it were the affected one. To ensure that the participants focused on the reflection, the unaffected arm was placed in the mirror box, and vision of the affected arm was occluded by a vertical board placed beside the mirror box. The activities consisted of transitive (eg, gross motor tasks, such as reaching
  Arms: Mirror Therapy

SUMMARY:
Stroke is a global health issue as this happens when the blood flow to the brain is disrupted or reduced, depriving the brain tissue of sugar and oxygen. This interruption affects the brain cells hence leading to the loss of a cell Various physical, cognitive and emotional losses are experienced. Cerebrovascular accident or simply stroke, is the fifth cause of mortality and one of the most common causes of disability in the United States of America (Campbell et al., 2019). There are two main types of stroke: ischemic and hemorrhagic. An ischemic stroke is characterized by an occlusion of a cerebral artery by an embolus or thrombus while hemorrhagic stroke results from a hemorrhage in the brain due to rupture of a blood vessel. A TIA or so-called mini stroke occurs when the clot is not severe enough to result in lasting symptoms (Feigin et al., 2022; Strilciuc et al., 2023).

Strokes substantially affect an individual mobility and overall quality of life, although few comparative studies comparing CIMT and MT exist in the literature. This research therefore seeks to systematically compare the effects of these two interventions on functional ambulation and quality of life of chronic stroke patients. Hereby, the research compares structured, task specific CIMT with the less structured, more general approach of MT in order to offer clinicians empirically founded recommendations on what course of action might prove effective for patients. This study also provides new insights to the field given that it not only describes the potential of CIMT within outpatient physiotherapy treatment but also provides an overview of the long-term effects for patients with stroke. These outcomes of this study will be useful in developing rehabilitative research, improving clinical practice protocols, and thereby improve the lifestyles of people living with chronic stroke.

DETAILED DESCRIPTION:
To compare the effects of MT and CIMT on functional ambulation and quality of life in chronic stroke patients.

Study Design: This was a randomized controlled trial with two parallel groups:

1. Group A (Constraint-Induced Movement Therapy (CIMT)):

   A well-defined and structured rehabilitation program that restricts the use of the unaffected limb to promote the functional recovery of the affected limb in chronic stroke patients(Franck et al., 2019).
2. Group B (Mirror Therapy):

A specific intervention that uses a mirror to create a visual illusion of the affected limb, with the goal of improving motor function and quality of life in chronic stroke patients

* Screening: Patients was screened to meet inclusion criteria. The consent form was taken from patients then patients was randomly allocated into two groups (33 in each group).
* Randomization: Patients fulfilling the inclusion criteria will be randomly divided into experimental and control groups using the computer software.
* Blinding: The study will be single blinded. The assessor, who has 5 years of experience in both clinical practice and research, will be unaware of the treatment given to both groups and will assess the participants objectively.
* Allocation: Allocation of the participants will be concealed, and envelope concealment method will be used for it.
* Outcome Measures:
* Functional Ambulation Categories (FAC)
* Tinetti gait and balance score (POMA)
* Short Form Health Survey (SF-12) Ethical Considerations: This study has received ethical approval from the Institutional Review Board (IRB). Informed consent was obtained from all participants.

Data Analysis: Statistical software was used to analyze the data, with appropriate tests employed based on data normality to compare outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants having age between 21 and 70 years old were recruited (e Silva et al., 2017).
* Both genders included (e Silva et al., 2017).

  * Diagnosed with post chronic hemiplegia ischemic stroke (≥6 months) affecting one side of the body(Danlami & Abdullahi, 2017; Mansfield et al., 2018).
* Participants having ability to follow verbal and visual instructions(Danlami & Abdullahi, 2017).
* Participants having no significant cognitive impairment (Minimental state examination score ≥ 17(Danlami & Abdullahi, 2017).
* Participants having low risk of fall (Tinetti gait and balance score ≥20)(Danlami & Abdullahi, 2017).

Exclusion Criteria:

* History of other neurological conditions affecting mobility. (Mansfield et al., 2018).
* Unstable fracture or other orthopedic conditions affecting gait such as OA, fracture and arthritis (Page et al., 2007).

  --Severe cognitive impairment.
* Participants with severe hemiparesis who are unable to reproduce movements accurately with the affected limb, as this may hinder active participation in the therapy(Danlami & Abdullahi, 2017; Ezendam et al., 2009).
* Individuals with physical limitations that prevent them from positioning themselves adequately to view their affected limb in the mirror during therapy sessions, as this could compromise the effectiveness of mirror therapy(Danlami & Abdullahi, 2017).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Categories (FAC) | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  Functional Ambulation Categories (FAC) is a 6-point functional walking test that provides the quantitative measurement of ambulation ability, which means how much human assistance the patient needs while walking, even with personal dual assistive device
Tinetti gait and balance score (POMA) | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  Tinetti Balance and Gait Assessment Performance Oriented Mobility Assessment (POMA) is a tool designed to assess the balance and gait status of a person with special reference to the potential for falling (Miodonska et al., 2018).
  . Scores are interpreted to reflect fall risk: Pollock et al. categories the serve self-tested mobility at low risk for participants scoring 25-28 points, moderate risk if scoring 19-24 points and high risk if scoring below 19 points on the scale. Also, patients with a score of below 26 are normally classified as high risk of falling.
Short Form Health Survey (SF-12) | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  The SF-12 scoring system generates two summary measures: th.e fact that the patients' disabilities are measured by the Physical Component Summary (PCS) and the Mental Component Summary (MCS). These scores are normalized based on a mean of 50 and standard deviation of 10 to obatain meaningful numerical values. Higher numbers represent better health related quality and those utilities with values above 50 represent superior health while below 50 represent inferior health. (Sampogna et al., 2019).

CONTACTS AND LOCATIONS:
Overall Officials: IQRA Mubeen, MS IN NEUROLOGY, Principal Investigator — University of Lahore; Asim Rana, MS MSK, Study Director — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezendam D, Bongers RM, Jannink MJ. Systematic review of the effectiveness of mirror therapy in upper extremity function. Disabil Rehabil. 2009;31(26):2135-49. doi: 10.3109/09638280902887768. PMID 19903124
- [Background] Iliyasu Z, Galadanci HS, Danlami KM, Salihu HM, Aliyu MH. Correlates of Postpartum Sexual Activity and Contraceptive Use in Kano, Northern Nigeria. Afr J Reprod Health. 2018 Mar;22(1):103-112. doi: 10.29063/ajrh2018/v22i1.10. PMID 29777647
- [Background] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727
- [Background] Campbell BCV, De Silva DA, Macleod MR, Coutts SB, Schwamm LH, Davis SM, Donnan GA. Ischaemic stroke. Nat Rev Dis Primers. 2019 Oct 10;5(1):70. doi: 10.1038/s41572-019-0118-8. PMID 31601801
- [Background] Rubiera M, Aires A, Antonenko K, Lemeret S, Nolte CH, Putaala J, Schnabel RB, Tuladhar AM, Werring DJ, Zeraatkar D, Paciaroni M. European Stroke Organisation (ESO) guideline on screening for subclinical atrial fibrillation after stroke or transient ischaemic attack of undetermined origin. Eur Stroke J. 2022 Sep;7(3):VI. doi: 10.1177/23969873221099478. Epub 2022 Jun 3. PMID 36082257